CLINICAL TRIAL: NCT04677426
Title: 129Xe Gas Exchange Imaging in IPF and cHP: A Reliability Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew Funding
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Duke University (Other); Children's Hospital Medical Center, Cincinnati (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00146495
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Hypersensitivity Pneumonitis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Alveolitis, Extrinsic Allergic | interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Progressive Interstitial Lung Disease (Experimental): Assess the intra-visit reliability and sensitivity to progression of 129Xe MR imaging measurements using a standardized imaging protocol in subjects with IPF and cHP.
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — Whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to assess patients with cHP and IPF.
  Other Names: Xenon; HP 129Xe

SUMMARY:
This research is a study to test the reliability of Hyperpolarized Xenon MRI (HXe MRI) as a biomarker in interstitial lung disease. The study is a non-randomized study to evaluate the test-retest performance of HXe MRI in Idiopathic Pulmonary Fibrosis (IPF) and chronic Hypersensitivity Pneumonitis (cHP) as a non-invasive biomarker of disease severity and prognosis. The study will include approximately 15 subjects with IPF, 15 subjects with cHP and 10 sex and age-matched normal controls performed across 3 sites.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Diagnosis of progressive chronic HP, IPF as determined by MDD discussion (historical or during screening period) OR normal control (no history of known lung disease, no abnormal parenchymal or airway findings on CT examination and no values outside of the normal for FVC, FEV1, TLC, and DLCO.)
* FVC % Predicted >45%
* DLCO % Predicted >30%
* Progressive lung disease as defined by one of the following criteria within 24 months of screening visit
* Relative decline in the FVC ≥ 10% of the predicted value
* Relative decline in the FVC of ≥ 5% - < 10% of the predicted value and worsening of respiratory symptoms
* Relative decline in the FVC of ≥ 5% - < 10% of the predicted value and an increased extent of fibrosis on prior clinical high-resolution CT
* Worsening of respiratory symptoms and an increased extent of fibrosis on high-resolution CT.

Exclusion Criteria:

* Stable FVC over 2-year period as determined by study physician
* Unstable cardiac condition within 6 months of screening as determined by study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
RBC:Barrier Ratio | RBC:Barrier will be assessed at Baseline and at 6 months.
  RBC:Barrier ratio will be determined using 129 Xenon MRI in 2 successive scans on two separate days 6 months apart. Same-day Repeated measures will be used to assess reliability of RBC:Barrier. Data acquired at 6 months will be correlated with FVC.

IPD SHARING:
Plan to Share IPD: No